CLINICAL TRIAL: NCT04400292
Title: Does the Concept of the Sentinel Lymph Node Apply to Esophageal Cancer? A Prospective Assessment of Near-infrared Image-guided Lymphatic Mapping and Sentinel Lymph Node Identification in Esophageal Cancer
Brief Title: Sentinel Lymph Node Mapping in Esophageal Cancer Using ICG Dye and NIR Imaging
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-201
Record Dates: First submitted 2020-05-20; First posted 2020-05-22 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Esophageal Cancer
Keywords: Sentinel Lymph Node Mapping; lymphadenectomy; esophagectomy; ICG Injection; Intraoperative NIR Imaging; 20-201
MeSH Terms: conditions — Esophageal Neoplasms | interventions — sarcolipin

STUDY DESIGN:
Intervention Model Description: This will be a prospective single-arm study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SLN mapping by NIR with ICG (Experimental): Patients will undergo ICG injection and NIR imaging for lymphatic mapping. Any identified SLNs will be dissected during the standard completion lymphadenectomy and esophagectomy. The SLN biopsy procedure will be performed as described below. Although NIR with ICG is used to assess conduit perfusion in all esophagectomies performed at MSK, its use for lymphatic mapping is considered experimental in esophageal cancer.
  Interventions: Other: Injection of indocyanine green (ICG)dye; Device: Near-Infrared Image-Guided; Procedure: Sentinel Lymph Node (SLN) mapping

INTERVENTIONS:
Other: Injection of indocyanine green (ICG)dye — Patients will receive a perilesional injection of indocyanine green (ICG) before the laparoscopic phase of the esophagectomy.
Device: Near-Infrared Image-Guided — Real-time near-infrared (NIR) fluorescence imaging will be performed by use of the Novadaq PINPOINT minimally invasive system with a laparoscopic camera.
Procedure: Sentinel Lymph Node (SLN) mapping — Any identified SLNs will be dissected during the standard completion lymphadenectomy and esophagectomy.

SUMMARY:
The purpose of this study is to find out whether sentinel lymph node (SLN) mapping with ICG dye and NIR imaging can be used to identify esophageal or esophagogastric junction cancer that has spread to the lymph nodes. If SLN mapping is successful in these types of cancer, surgeons in the future could identify the sentinel lymph nodes and only remove these instead of removing all the lymph nodes which is currently done.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of adenocarcinoma tumor located in distal 1/3 of esophagus or esophagogastric junction , with a plan to undergo minimally invasive esophagectomy.
* All patients with Stage IVA (AJCC Cancer Staging Manual, 8th edition) disease will be eligible
* ≥18 years of age.
* Documented, signed, and dated informed consent, obtained before any procedures, for the proposed research study and for standard surgical resection.

Exclusion Criteria:

* No plan to undergo surgical resection.
* Severe iodide or seafood allergy.
* Women of childbearing potential without a negative pregnancy test; or women who are lactating.
* Prior diagnosis of severe hepatic or renal dysfunction.
* Patients with Stage IVB or M1 disease (AJCC Cancer Staging Manual, 8th edition)
* Patients with local recurrence and planning to undergo salvage esophagectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The number of lymph nodes visualized to be fluorescent and nonfluorescent. | 1 year
  Surgical data will include the number of lymph nodes identified and removed both NIRfluorescent and NIR-nonfluorescent nodes.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Molena, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm